CLINICAL TRIAL: NCT07074977
Title: An Exploratory Proof of Concept Study to Assess the Pharmacokinetics/Pharmacodynamics (PK/PD) of Nemolizumab in Adult Participants With Chronic Pruritus of Unknown Origin (CPUO)
Brief Title: Proof of Concept Study to Assess the Pharmacokinetics/Pharmacodynamics of Nemolizumab in Adults With Chronic Pruritus of Unknown Origin (CPUO)
Acronym: CPUO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPR207913
Record Dates: First submitted 2025-06-24; First posted 2025-07-20 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pruritus of Unknown Origin
MeSH Terms: interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- nemolizumab (Experimental): Participants weighing < 90 kg will receive one subcutaneous (SC) injection of 30 milligrams (mg) nemolizumab (with 60 mg loading dose at baseline) every 4 weeks (Q4W) at Weeks 4, 8, and 12. Participants weighing >= 90 kg will receive two SC injections of 30 mg nemolizumab ( 60 mg total) at baseline (without loading dose) and at Weeks 4, 8, and 12.
  Interventions: Drug: nemolizumab
- Placebo (Placebo Comparator): Participants weighing < 90 kg will receive two SC injections of matching placebo at baseline followed by 1 SC injection Q4W at Weeks 4, 8 and 12. Participants weighing >= 90 kg will receive two SC injections of matching placebo at baseline and at Weeks 4, 8, and 12.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: nemolizumab — Participants will receive either 30 mg or 60 mg dose of nemolizumab as SC injection.
  Other Names: CD14152
  Arms: nemolizumab
Drug: Placebo — Participants will receive matching placebo as SC injection.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the PK/PD relationship of nemolizumab in adult participants aged 18 years or above with chronic pruritus of unknown origin (CPUO) during a 16-week treatment period.

DETAILED DESCRIPTION:
This study is to assess the PK/PD relationship of nemolizumab in adult participants with CPUO. The study will consist of a 2 to 4-week screening period, a 16-week treatment period, and an 8-week follow up period (12 weeks after last study drug injection). Participants will be randomized 4:1 to nemolizumab or placebo. Dosing will be adjusted according to participants body weight ( less than [<] 90 kilograms [kg] versus >= 90 kg). Participation in the study will last up to 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:

  1. Participant must be 18 years of age or older.
  2. Participants with chronic pruritus on normal-appearing skin (except for dry skin or excoriations) for at least 6 months before the screening visit.
  3. Chronic pruritus considered of unknown origin (i.e., without a clear association to another condition or medication) as assessed by the investigator at baseline.
  4. The pruritus must affect at least 4 of the following body areas: left lower limb, right lower limb, left upper limb, right upper limb, anterior trunk, posterior trunk.
  5. History of insufficient control of the chronic pruritus with prior treatment.
  6. Peak Pruritus Numeric Rating Scale (PP NRS) score greater than and equal to (>=) 7 in the 24-hour period prior to the Screening visit.
  7. Weekly average Peak Pruritus Numeric Rating Scale (PP NRS) score >= 7 in the week (7 days) immediately prior to randomization, as recorded in the patient diary.
  8. Female of childbearing potential must agree to use at least 1 adequate and approved method of contraception throughout the study and for 12 weeks after the last study intervention injection.

     Contraceptive use by participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
  9. Females of non-childbearing potential must meet 1 of the following criteria:
* Absence of menstrual bleeding for 1 year prior to screening without any other medical reason, confirmed with follicle stimulating hormone (FSH) level in the postmenopausal range
* Documented hysterectomy, bilateral salpingectomy, or bilateral oophorectomy at least 3 months before screening 10. Signed informed consent. 11. Participant is willing and able to comply with all of the time commitments and procedural requirements of the clinical study protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply :

Medical Conditions

1. Known dermatologic, systemic, neurologic or psychiatric condition(s), other than dry skin, that considered by the investigator to be the primary cause of current pruritus.
2. Documented parasitic infection, including skin parasites such as scabies, within 12 weeks prior randomization.
3. Cutaneous infection within 1 week before the baseline visit, any infection requiring treatment with oral or parenteral antibiotics, antivirals, antiparasitics, or antifungals within 2 weeks before the baseline visit.
4. Diagnosis of chronic pruritus of neuropathic origin including but not limited to scalp dysesthesia, brachioradial pruritus, generalized neuropathic pruritus or chronic pruritus of psychogenic origin (pruritus associated with psychological disorders such as delusional parasitosis or Morgellons disease).
5. Any medical or psychological condition or any clinically relevant laboratory abnormalities that put the participant at significant risk.
6. History of bullous pemphigoid or positive bullous pemphigoid autoantibodies at screening.
7. History of mastocytosis or serum total tryptase greater than (>) 20 nanograms per milliliter (ng/ml) at screening.
8. Active tuberculosis (TB) or non-tuberculosis mycobacterial infection, or a history of incompletely treated TB.
9. Positive serology results Hepatitis B surface antigen or (HBsAg) or Antibody to Hepatitis B core antigen (HBcAb), Hepatitis C virus (HCV) antibody with positive confirmatory test for HCV (e.g., polymerase chain reaction [PCR]), or Human Immunodeficiency Virus [HIV] antibody) at the screening visit.
10. Known or suspected immunodeficiency.
11. Lymphoproliferative disease or malignancy within the last 5 years.
12. Presence of major psychiatric diagnosis, clinically significant dementia, intellectual impairment, or any medical condition or disability which, in the investigator's opinion, may confound the assessment of nemolizumab's safety or efficacy or interfere with the participant's ability to comply with protocol mandated activities.
13. Receipt of prohibited medications within the specified timeframe before the baseline visit
14. Previous participation in a clinical study with nemolizumab
15. Currently participating or participated in any other study of an investigational drug or device, within the past 8 weeks (or 5 half-lives of the investigational drug, whichever is longer) before the screening visit, or is in an exclusion period (if verifiable) from a previous study.
16. Body weight < 30 kg.
17. Prior treatment with commercially available nemolizmab
18. Hypersensitivity to the active substance (nemolizumab) or to any of the excipients of the study intervention.
19. Requiring rescue therapy for pruritus during the screening period.
20. Alcohol or substance abuse within 6 months of the screening visit.
21. Planned or anticipated major surgical procedure or other activity that would interfere with the participant's ability to comply with protocol-mandated assessments.
22. Pregnant or breastfeeding female, or female planning a pregnancy during the study.
23. Vulnerable participant as defined by International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Population Pharmacokinetics (PopPK) Model of the Elimination of nemolizumab During the 16-week Treatment Period Point | From Baseline up to Week 16
  Point Estimate of Population Total Clearance (Cl/F) of nemolizumab will be reported.
Population Pharmacokinetics (PopPK) Model of the Distribution of nemolizumab During the 16-week Treatment Period Point | From Baseline up to Week 16
  Point Estimate of Population Volume of Distribution (Vd/F) of nemolizumab will be reported.
Population Pharmacokinetics (PopPK) Model of the Absorption of nemolizumab During the 16-week Treatment Period Point | From Baseline up to Week 16
  Point Estimate of Absorption Rate Constant (Ka) of nemolizumab will be reported.
Pharmacokinetic (PK)/Pharmacodynamic (PD) Model of the Effect of nemolizumab Systemic Exposure on Pruritus during 16-week Treatment Period | From Baseline up to Week 16
  Point Estimate of population IC50 of nemolizumab, i.e. the drug concentration required to produce 50% of the maximal inhibition of Average Peak Pruritus, will be reported.

SECONDARY OUTCOMES:
Individual Observed Ctrough Concentrations of nemolizumab | Week 16
  Average of individual observed Ctrough concentrations of nemolizumab at week 16 will be reported.
Individual Model - derived Ctrough Concentrations of nemolizumab | Week 16
  Average of individual model-derived Ctrough concentrations of nemolizumab at week 16 will be reported.
Individual Total Clearance (Cl/F) of nemolizumab | From Baseline up to Week 16
  Average of individual model-derived estimates of Cl/F will be reported.
Individual Volume of Distribution (Vd/F) of nemolizumab | From Baseline up to Week 16
  Average of individual model-derived estimates of Vd/F will be reported.
Individual Absorption Rate Constant (Ka) of nemolizumab | From Baseline up to Week 16
  Average of individual model-derived estimates of Ka will be reported.
Individual Maximum Serum Concentration (Cmax) of nemolizumab | From Baseline up to Week 16
  Average of individual model-derived estimates of Cmax will be reported.
Individual Time to Reach Maximum Serum Concentration (Tmax) of nemolizumab | From Baseline up to Week 16
  Average of individual model-derived estimates of Tmax will be reported.
Individual Area Under the Concentration-time Curve Within a Dosing Interval (AUCtau) of nemolizumab | From Baseline up to Week 16
  Average of individual model-derived estimates of AUCtau will be reported.
Terminal Half-life (t1/2) of nemolizumab | From Baseline up to Week 16
  Average of individual model-derived estimates of t1/2 will be reported.
Change From Baseline in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) | Up to Week 16
  PP NRS is a scale that will be used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores are provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome. Participant will report PP NRS via daily e-PRO diary.
Number of Participants With Adverse Events (AEs), Treatment Emergent Adverse Events (TEAEs), Adverse Events of Special Interest (AESIs), and Serious Adverse Events (SAEs), AEs Leading to Study Intervention Withdrawal, AEs Leading to Study Discontinuation | From start of study up to follow-up period (Week 24)
  AE defined as any untoward medical occurrence in clinical study participant administered a medicinal product which does not necessarily have causal relationship with this treatment. TEAEs defined as AEs occurring after first administration of study drug during the study. SAE was any untoward medical occurrence, in view of either Investigator or Sponsor, that resulted in death, was life-threatening, resulted in inpatient hospitalisation or prolongation of existing hospitalisation, resulted in persistent or significant disability/incapacity, was congenital anomaly/birth defect or was important medical event. AESI was noteworthy TEAE for study drug that was to be monitored closely and reported promptly. Relatedness to study drug was based on Investigator's discretion. AEs Leading to study treatment withdrawal and AEs Leading to study withdrawal will also be reported.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Galderma Investigational Site (site# 8893), Birmingham, Alabama
  - Galderma Investigational Site (site# 8130), Los Angeles, California
  - Galderma Investigational Site (site# 8021), San Diego, California
  - Galderma Investigational Site (site# 7075), San Francisco, California
  - Galderma Investigational Site (site# 7054), Tampa, Florida
  - Galderma Investigational Site (site# 8142), Indianapolis, Indiana
  - Galderma Investigational Site (site# 8743), Ann Arbor, Michigan
  - Galderma Investigational Site (site# 8521), Saint Joseph, Missouri
  - Galderma Investigational Site (site# 8108), Las Vegas, Nevada
  - Galderma Investigational Site (site# 7110), New City, New York
  - Galderma Investigational Site (site# 7111), Fargo, North Dakota
  - Galderma Investigational Site (site# 8003), Webster, Texas
  - Galderma Investigational Site (site# 8862), Fairfax, Virginia
  - Galderma Investigational Site (site# 8725), Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No